CLINICAL TRIAL: NCT05466461
Title: Clinical Assessment of Injectable Flowable Composite With Giomer Based Technology Versus Smart Bioactive Restoration in Carious Class V Cavities (A Randomized Clinical Trial)
Brief Title: Clinical Assessment of Giomer Based Technology Versus Smart Bioactive Restoration in Carious Class V Cavities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Bassma Reda Abdelhafeez, Principle Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 236756
Record Dates: First submitted 2022-07-15; First posted 2022-07-20 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries | interventions — ACTIVA BioACTIVE-RESTORATIVE

STUDY DESIGN:
Intervention Model Description: Compare between S-PRG-containing injectable flowable resin composite (Beautifil Flow Plus X) and smart bioactive flowable resin composite (Activa bioactive restorative) over one year through evaluation of the modified USPHS clinical performance in patients with carious class V moderately deep cavities.
Who Masked: Participant, Outcomes Assessor
Masking Description: During treatment, the type of material will be concealed from the patient, and the patient will have no information which material will be used. The type of restoration will not mentioned in the patient's file. Instead, it will be replaced by a combination which the evaluators will be not familiar with. The operator will be blinded for the type of restoration during tooth preparation and was informed only at the time of restoration placement. The purpose of this discretion is to ensure double blinding both at the patient, as well as the evaluators level.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Beautifil Flow Plus X. (Experimental): Giomers is a hybrid material category which contains Surface Pre-Reacted Glass-ionomer filler or S-PRG filler is produced from fluoroboro-alumino-silicate glass and polyacrylic acid through an acid-base reaction to form a stable glass ionomer phase on glass filler particle surfaces. S-PRG fillers can release and recharge fluoride. Also, the S-PRG filler-containing resinous materials are able to release various ions, such as aluminum (Al3+), boron (BO3 3-), fluoride (F- ), sodium (Na+), silicon (SiO3 2-), and strontium (Sr2+), in neutral and acidic conditions.
  Interventions: Procedure: Beautifil Flow Plus X.
- Activa bioactive restorative (Active Comparator): Activa BioACTIVE Restorative (Activa), developed by Pulpdent (Watertown, MA, USA), is a new bioactive restorative material that combines the advantages of an RMGIC (resin modified glass ionomer cement) and RBC (resin based composite), representing a new category of restorative materials that are ion releasing. It contains methacrylate- based monomers, a modified polyacrylic acid, modified Diurethane Dimethacrylate (rubberized resin), and fillers
  Interventions: Procedure: Activa bioactive restorative

INTERVENTIONS:
Procedure: Beautifil Flow Plus X. — Class V cavities will be prepared, Selective etching technique will be used with phosphoric acid etching gel for 15 seconds on enamel.Single Bond TM Universal will be applied to cavity walls and margins with agitation for 20 seconds.The adhesive will be light-cured for 20 seconds. Then Beautifil Flow Plus X composite will be placed
  Arms: Beautifil Flow Plus X.
Procedure: Activa bioactive restorative — Class V cavities will be prepared, Selective etching technique will be used with phosphoric acid etching gel for 15 seconds on enamel. Bonding agent will be applied on the entire cavity and light-cured for 20 seconds then Activa bioactive restorative composite will be applied and cured for 20 seconds.
  Arms: Activa bioactive restorative

SUMMARY:
This study will compare between S-PRG-containing injectable flowable resin composite (Beautifil Flow Plus X) and smart bioactive flowable resin composite (Activa bioactive restorative) through evaluation of the modified USPHS clinical performance in patients with carious class V moderately deep cavities.

DETAILED DESCRIPTION:
Bioactive glass has an amorphous structure, whereas glass-ceramics are crystallized glasses and composites of a crystalline phase in a residual glassy phase. Bioactive glass consists solely of the elements found in the body material, mainly being silicon (Si), calcium (Ca), sodium (Na), phosphorous (P), and oxygen (O) . Among the diverse kinds of bioactive glass filler, surface pre- reacted glass ionomer (S-PRG) filler has already been used for a relatively long time in some specific commercial RBCs. Most studies investigating this material assortment have focused on ion-release degree and potentially associated antibacterial effects. The restoration's surface integrity may be a key factor determining the eventual clinical beneficial effect of the alleged antibacterial properties. The antibacterial efficacy of bioactive glass depends on the concentration of the ions released from the glass.

As inorganic bioactive fillers, S-PRGs have the additional ability to release ions. S-PRG filler is considered a multifunctional bioactive glass because it can release several types of ions including Al, B, F, Na, Si, and Sr. The released ions can exhibit a variety of bioactive behaviors, such as preventing fungal and bacterial adhesion, antibacterial activity, neutralizing acids, inhibiting demineralization, and enhancing remineralization.

The biological effects of S-PRG fillers have been studied for several types of oral pathogens. It was reported that the elute of the S-PRG filler has a protective effect against Streptococcus mutans. Moreover, the elute of S-PRG filler reduced the density and thickness of the formed biofilm.

ELIGIBILITY:
Inclusion Criteria:

* ages 18 to 55 years.
* Male or female patients.
* Patients with no history of allergic reactions to methacrylate compounds and in good general health.
* Patients with good general health.
* Patients with good recall availability. Patients required Class V restoration
* Vital teeth with normal appearance and morphology.
* Absence of clinical symptoms of irreversible pulpitis, such as spontaneous pain or sensitivity to pressure.
* Absence of clinical diagnosis of pulp exposure, fistula, swelling of periodontal tissues, and/or abnormal tooth mobility .
* No defects and lesions for other operative intervention, occlusal and proximal contacts with adjacent teeth.

Exclusion Criteria:

* Patients with history of any adverse reaction to clinical materials of the types to be used in the evaluation.

  * Pregnant and lactating females.
  * Any patients with medical and/or dental histories which could possibly complicate the provision of the proposed restoration and/or influence behavior and performance of the restorations in clinical service.
  * They are included in the evaluation of other restorative materials and systems involving the anterior and/or posterior teeth.
  * Patients who maintain an unacceptable standard of oral hygiene.
  * Teeth with noncarious cervical lesions.
  * Severe tooth sensitivity.
  * Non-vital or fracture or cracked teeth.
  * Tooth with defective restoration.
  * Teeth with advanced periodontal diseases.
  * There is evidence occlusal parafunctions and/or atypical tooth wear.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Assessment of Modified USPHS Criteria (Marginal discoloration) change over time | Change between baseline,6 months and 12 months
  Alfa: there is no visual evidence of marginal discoloration different from the color of the restorative material and from the color of the adjacent tooth structure.
  Bravo: there is visual evidence of marginal discoloration at the junction of the tooth structure and the restoration that has not penetrated along the restoration in a pulpal direction.
  Charlie: there is visual evidence of marginal discoloration at the junction of the tooth structure and the restoration, but the discoloration has penetrated along the restoration in a pulpal direction.

SECONDARY OUTCOMES:
Assessment of Modified USPHS criteria. (Secondary caries) change over time | Change between baseline,6 months and 12 months
  Alfa: no caries is present. Charlie: caries is present.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

REFERENCES:
- [Background] Yoshihara K, Nagaoka N, Maruo Y, Sano H, Yoshida Y, Van Meerbeek B. Bacterial adhesion not inhibited by ion-releasing bioactive glass filler. Dent Mater. 2017 Jun;33(6):723-734. doi: 10.1016/j.dental.2017.04.002. Epub 2017 Apr 29. PMID 28465066
- [Background] Nomura R, Morita Y, Matayoshi S, Nakano K. Inhibitory effect of surface pre-reacted glass-ionomer (S-PRG) eluate against adhesion and colonization by Streptococcus mutans. Sci Rep. 2018 Mar 22;8(1):5056. doi: 10.1038/s41598-018-23354-x. PMID 29568011
- [Background] Tonprasong W, Inokoshi M, Tamura M, Uo M, Wada T, Takahashi R, Hatano K, Shimizubata M, Minakuchi S. Tissue Conditioner Incorporating a Nano-Sized Surface Pre-Reacted Glass-Ionomer (S-PRG) Filler. Materials (Basel). 2021 Nov 4;14(21):6648. doi: 10.3390/ma14216648. PMID 34772173